CLINICAL TRIAL: NCT01860755
Title: Physiotherapy Treatment (Including Vestibular Rehabilitation) Compared to Rest in Individuals With Persistent Symptoms of Dizziness, Neck Pain and/or Headache Following Sport-related Concussion.
Brief Title: Effects of Physiotherapy in Individuals With Persistent Symptoms Following Concussion
Acronym: PTConc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sport Injury Prevention Research Centre (Other)
Collaborators: Alberta Centre for Child, Family & Community Research (Other); University of Calgary (Other); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SIPRC-PT-conc-01
Record Dates: First submitted 2013-05-20; First posted 2013-05-23 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Sport-related Concussion
Keywords: Sport-related concussion; Dizziness; Neck pain; Headaches; Physiotherapy; Treatment
MeSH Terms: conditions — Dizziness; Neck Pain; Headache | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy (Experimental): Physiotherapy: including vestibular rehabilitation and multimodal treatment for the cervical spine, once weekly with the study physiotherapist for 8 weeks or until time of medical clearance to return to sport. This group also received the control intervention.
  Interventions: Other: Control postural education, general range of motion and strengthening in addition to the standard of care; Other: Physiotherapy
- Control (Active Comparator): Control: postural education, general range of motion and strengthening in addition to the standard of care rest followed by graded exertion. Individuals were seen once weekly for eight weeks or until time of medical clearance to return to sport.
  Interventions: Other: Control postural education, general range of motion and strengthening in addition to the standard of care

INTERVENTIONS:
Other: Control postural education, general range of motion and strengthening in addition to the standard of care — Control: postural education, general range of motion and strengthening in addition to the standard of care rest followed by graded exertion. Individuals were seen once weekly for eight weeks or until time of medical clearance to return to sport.
Other: Physiotherapy — Physiotherapy: including vestibular rehabilitation and multimodal treatment for the cervical spine, once weekly with the study physiotherapist for 8 weeks or until time of medical clearance to return to sport.
  Arms: Physiotherapy

SUMMARY:
The purpose of this study is to determine the effects of a combined physiotherapy treatment (including vestibular rehabilitation and treatment for the cervical spine) in youth and young adults with ongoing symptoms of dizziness, neck pain and headaches following a sport-related concussion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Sport-related concussion as per the Third International Consensus Guidelines
* Persistent symptoms (greater than 10 days) of dizziness, unsteadiness, neck pain and/or headaches reported on the Sport Concussion Assessment Tool 2 (SCAT2)
* Clinical examination findings suggesting vestibular and/or cervical spine involvement

Exclusion Criteria:

* Fracture, other neurological conditions, musculoskeletal injuries (other than the cervical spine) that restrict activity and medications that affect neural adaptation

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Days to medical clearance to return to sport | up to 8 weeks
  Number of days to medical clearance by study physician

SECONDARY OUTCOMES:
Change in Numeric Pain Rating Scale Score-Neck Pain | Change between Baseline and 8 weeks or time of medical clearance
  Self-reported cervical spine pain rated on a scale of 0-10
Change in Numeric Dizziness rating Score | Change between Baseline and 8 weeks or time of medical clearance
  Self reported dizziness on a scale of 0-10
Change in Numeric Pain Rating Scale Score-Headache | Change between Baseline and 8 weeks or at time of medical clearance
  Self-report score for headache on a scale of 0-10
Change in Activities Specific Balance Confidence Scale Score | Change between Baseline and 8 weeks or time of medical clearance
  Self report measure of confidence during 16 balance activities
Change in Dizziness Handicap Index Score | Change between Baseline and 8 weeks or time of medical clearance
  Self report measure evaluating perceived handicap secondary to dizziness
Change in Sport Concussion Assessment Tool 2 (SCAT2) | Change between Baseline and 8 weeks or time of medical clearance
  Multifaceted tool used in the assessment of concussion and includes domains of symptom report, cognitive function, balance and coordination
Change in Dynamic Visual Acuity | Change between Baseline and 8 weeks or time of medical clearance
  Assessed clinically using an eye chart and a metronome set at 2 Hz. Static visual acuity is measured 13 feet from the target. The subjects head is rotated at 2 Hz and visual acuity is measured dynamically. The difference between static and dynamic visual acuity is calculated.
Head Thrust Test | Baseline and at 8 weeks or time of medical clearance
  Clinical test performed in sitting with head flexed and high velocity low amplitude motion into 5-15 degrees rotation is performed while the subject is asked to maintain focus with the examiner's nose.
Change in modified Motion Sensitivity Test Score | Change between Baseline and 8 weeks or time of medical clearance
  Patient report of intensity and duration of dizziness with eight head or body motions
Change in Functional Gait Assessment Score | Change between Baseline and 8 weeks or time of medical clearance
  Dynamic Balance Measure that includes 10 different movements and the ability to complete each activity is rated by the examiner.
Change in Cervical Flexor Endurance | Change between Baseline and 8 weeks or time of medical clearance
  Test to evaluate the time (seconds) that an individual can maintain the head in a position of craniovertebral flexion and two finger widths above a pillow in crook lying.
Change in Joint Position Error | Change between Baseline and 8 weeks or time of medical clearance
  Clinical test using a laser pointer affixed to a head piece on top of the head that is projected onto a bull's eye target. Subject rotates head to left, right (rotation) or up (extension) to the maximum comfortable range and relocates to the perceived point of neutral head position with eyes closed. A measures from the centre of the bull's eye is recorded. A mean of three trials is recorded for each direction.

CONTACTS AND LOCATIONS:
Overall Officials: Willem H Meeuwisse, MD, PhD, Principal Investigator — Sport Injury Prevention Research Centre, University of Calgary; Carolyn A Emery, PT, PhD, Principal Investigator — Sport Injury Prevention Research Centre, University of Calgary; Kathryn J Schneider, PT, PhD, Study Director — Sport Injury Prevention Research Centre, University of Calgary
Locations (1):
- Sport Injury Prevention Research Centre, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Schneider KJ, Meeuwisse WH, Nettel-Aguirre A, Barlow K, Boyd L, Kang J, Emery CA. Cervicovestibular rehabilitation in sport-related concussion: a randomised controlled trial. Br J Sports Med. 2014 Sep;48(17):1294-8. doi: 10.1136/bjsports-2013-093267. Epub 2014 May 22. PMID 24855132